CLINICAL TRIAL: NCT00427427
Title: A Phase II Trial of Delayed Adjuvant Herceptin® in Patients With HER-2 Positive Breast Cancer
Brief Title: Delayed Adjuvant Herceptin® Treatment in Patients With HER-2 Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 06-05-104; H3754s
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2007-10

CONDITIONS: Breast Cancer
Keywords: non-metastatic breast cancer; HER-2 positive breast cancer; Herceptin (trastuzumab); delayed adjuvant therapy; acceptability rate; non-metastatic, HER-2 positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab

SUMMARY:
The purpose of the study is to determine what factors affect a patient's decision to accept delayed Herceptin® treatment after completing their surgery and/or chemotherapy and/or radiation therapy.

Women with invasive breast cancer that have a HER-2 positive (FISH +) determination in 2004 or thereafter and who have completed surgery and primary treatment earlier will be potentially eligible.

Patients will be asked to complete a questionnaire about their breast cancer and reasons why they may or may not accept Herceptin® treatment. Patients will be given the option to (1) receive Herceptin® for 52 weeks and have annual doctor visits for 5 years or (2) not to receive Herceptin® but agree to annual doctor visits for 5 years.

DETAILED DESCRIPTION:
Study Phase- Phase II Study Type- Interventional Study Design-

This is an open label, non-randomized phase II study in patients with non-metastatic HER-2 positive breast cancer by FISH diagnosed in 2004 or thereafter. Potential patients will sign a written ICF prior to completing a questionnaire designed to determine what factors may affect a patient's acceptance of Herceptin® treatment. After answering the questionnaire, patients will be given the following options:

1. to receive one year of trastuzumab treatment and annual follow-up for 5 years
2. to decline trastuzumab treatment but serve as a comparison group member for monitoring safety and effectiveness of trastuzumab and to have annual follow-up for 5 years

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed non-metastatic infiltrating carcinoma of the breast.
2. HER-2 amplified (FISH +) determination in 2004 or thereafter.
3. ECOG performance status 0-2.
4. Patients 18 years of age or older.
5. HER-2 status is determined by FISH test.
6. The following criteria are applicable to the trastuzumab treatment group:

   * Normal LVEF as determined by ECHO or MUGA. If baseline LVEF > 75%, then LVEF shall be repeated to determine if falsely elevated.
   * Adequate bone marrow function as indicated by the following: ANC >1500/mL, Platelets >/=100,000/mL, Hemoglobin >9 g/dL
   * Adequate renal function,as indicated by serum creatinine </= 1.5 x ULN
   * Adequate liver function, as indicated by total bilirubin </= 1.5 x ULN
   * AST and ALT < 2 x ULN unless related to primary disease.
   * If female of childbearing potential, pregnancy test (blood or urine) is negative and she agrees to use effective birth control method for the duration of the study.
7. Signed informed consent has been obtained.

Exclusion Criteria:

1. Non-confirmed HER-2 positive by FISH infiltrating carcinoma of the breast.
2. Evidence of metastatic disease.
3. Previous trastuzumab treatment.
4. Concurrent anticancer treatment other than hormonal agents (tamoxifen, aromatase inhibitors) or radiotherapy.
5. Patient with history of or active cardiac disease, including cardiomyopathy, congestive heart failure, prior myocardial infarction, or arrhythmia.
6. Symptomatic intrinsic lung disease resulting in dyspnea at rest.
7. Concurrent life-limiting disease with a life expectancy of less than one year.
8. Pregnancy, nursing women, and fertile women who do not practice birth control.
9. Inability to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To evaluate acceptance rate of delayed adjuvant trastuzumab treatment.
To evaluate signs and symptoms of cardiotoxicity.

SECONDARY OUTCOMES:
Annual assessment of recurrent disease.
Overall survival and disease specific survival.

CONTACTS AND LOCATIONS:
Overall Officials: Helena R Chang, M.D, Ph.D., Principal Investigator — Revlon/UCLA Breast Center
Locations (1):
- Revlon/UCLA Breast Center, Los Angeles, California, United States